CLINICAL TRIAL: NCT04050059
Title: Comparison of Two Analgesic Pretreatment Techniques (2% Lidocaine Infiltration vs. EMLA Cream Application) Before Spinal Needle Insertion for Pain Reduction and Maternal Satisfaction Level Assessment in Women Undergoing LSCS. A Prospective Randomized Control Trial
Brief Title: Comparison of Two Analgesic Pretreatment Techniques Before Spinal Needle Insertion for Pain Reduction and Maternal Satisfaction Level Assessment in Women Undergoing LSCS.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Dr. Malika Hameed, Fellow Obstetric Anesthesiology, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019-1791-4956
Record Dates: First submitted 2019-08-04; First posted 2019-08-08 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Anesthesia, Spinal; Pain; Pregnancy; Cesarean Section
MeSH Terms: conditions — Pain | interventions — Lidocaine, Prilocaine Drug Combination; Lidocaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2% Lidocaine group (Active Comparator): In 2% lidocaine group infiltration (Xylocaine 2% Barrett Hodgson Pakistan Pvt limited) skin and subcutaneous tissue will be infiltrated with 3 ml of 2% lidocaine (dose of 60 mg) before spinal anesthesia induction.
  Interventions: Drug: 2% lidocaine
- EMLA cream group (Active Comparator): In EMLA (Eutectic Mixture of Local Anesthesia- lidocaine 2.5% and prilocaine 2.5%) cream group, EMLA cream (5g tube Aspen pharma trading limited) will be applied topically in dose of 2.5 grams (half tube of cream) and area will be covered with tegaderm dressing. Application of EMLA will at least stay for 30 minutes before spinal needle insertion
  Interventions: Drug: EMLA cream

INTERVENTIONS:
Drug: EMLA cream — EMLA cream (5g tube Aspen pharma trading limited) will be applied topically in dose of 2.5 grams (half tube of cream) and area will be covered with tegaderm dressing. Application of EMLA will at least stay for 30 minutes before spinal needle insertion
  Arms: EMLA cream group
Drug: 2% lidocaine — In 2% lidocaine group infiltration (Xylocaine 2% Barrett Hodgson Pakistan Pvt limited), skin and subcutaneous tissue will be infiltrated with 3 ml of 2% lidocaine (dose of 60 mg) before spinal needle insertion
  Arms: 2% Lidocaine group

SUMMARY:
Nowadays lower segment cesarean sections are preferably carried out under regional anesthesia due to multiple advantages.

Local infiltration of lidocaine or any other anesthetic is used before lumber puncture in many centers to reduce needle stick pain.

EMLA (eutectic mixture of local anesthetic) cream is the combination of lidocaine and prilocaine which have been effectively used in few studies to reduce needle prick pain.

We would like to see which analgesic pretreatment is superior in terms of reducing pain of spinal needle insertion and have better maternal satisfaction levels.

DETAILED DESCRIPTION:
OBJECTIVES: To compare the pain reduction and maternal satisfaction levels of two analgesic pretreatment modalities on pain reduction of spinal needle insertion i.e. 2% lidocaine infiltration and EMLA in patients undergoing elective LSCS.

Hypothesis: Analgesic pre-treatment with EMLA is superior to local skin infiltration with lidocaine

ELIGIBILITY:
Inclusion Criteria:

* All adult women undergoing elective LSCS under spinal anesthesia

Exclusion Criteria:

* BMI of more than 35 kg/m2
* Contraindication to spinal anesthesia
* Spinal deformity
* Refusal of regional anesthesia
* Patients with a history of back surgery
* confirmed allergy to local anesthetics
* More than three attempts of needle insertion for inducing spinal anesthesia

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female pregnant patient planned for elective cesarean section under spinal anesthesia
Enrollment: 62 (Actual)
Dates: Start 2019-11-13 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
Pain Score (Subjective) | After 10 minutes (right after spinal anesthesia procedure is complete)
  Visual Analogue Scale pain Score in cm
Pain Score (Objective) | During spinal anesthesia procedure
  Objective scoring:
  1= No pain 2 = Mild flinch 3 = Wince 4= Yelp 5= Pulled away
Maternal Satisfaction | After 10 minutes (right after spinal anesthesia procedure is complete)
  Maternal Satisfaction Score (end of spinal anesthesia):
  Very Satisfied Satisfied No comments Unsatisfied Very Unsatisfied

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan

REFERENCES:
- [Background] Koscielniak-Nielsen Z, Hesselbjerg L, Brushoj J, Jensen MB, Pedersen HS. EMLA patch for spinal puncture. A comparison of EMLA patch with lignocaine infiltration and placebo patch. Anaesthesia. 1998 Dec;53(12):1218-22. doi: 10.1046/j.1365-2044.1998.00608.x. PMID 10193230
- [Background] Sharma SK, Gajraj NM, Sidawi JE, Lowe K. EMLA cream effectively reduces the pain of spinal needle insertion. Reg Anesth. 1996 Nov-Dec;21(6):561-4. PMID 8956393
- [Background] Wenk M, Massoth C, Weidlich S, Pöpping D M, Gurlit S, et al. Effects of local skin anaesthesia on pain during lumbar puncture. J Anaesthesiol Crit Care. 2017;1 (1):1-5
- [Background] Juarez Gimenez JC, Oliveras M, Hidalgo E, Cabanas MJ, Barroso C, Moraga FA, Gallego S, de Toledo JS. Anesthetic efficacy of eutectic prilocaine-lidocaine cream in pediatric oncology patients undergoing lumbar puncture. Ann Pharmacother. 1996 Nov;30(11):1235-7. doi: 10.1177/106002809603001104. PMID 8913402